CLINICAL TRIAL: NCT03450928
Title: Peroral Endoscopic Myotomy (POEM) for the Treatment of Esophageal Achalasia: Long vs Short Myotomy. Prospective Randomized Controlled Study
Brief Title: POEM: Long vs Short Myotomy for Achalasia. RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Guido Costamagna, Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POEMLvS
Record Dates: First submitted 2017-11-07; First posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Achalasia
Keywords: Peroral Endoscopic Myotomy; Endoscopy; POEM; Submucosal endoscopy
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short POEM (Active Comparator): Patients in the Short POEM-group will undergo a Peroral Endoscopic Myotomy (POEM) extended for a total of 7 cm (including 4 cm above the esophago-gastric junction and 3cm on the stomach).
  Interventions: Procedure: Peroral Endoscopic Myotomy (POEM)
- Long POEM (Active Comparator): Patients in the Long POEM-group will receive a 12cm-long Peroral Endoscopic Myotomy (POEM), including 9 cm on the esophagus and 3cm on the gastric wall
  Interventions: Procedure: Peroral Endoscopic Myotomy (POEM)

INTERVENTIONS:
Procedure: Peroral Endoscopic Myotomy (POEM) — Peroral endoscopic myotomy (POEM) is a minimally invasive intervention for the treatment of esophageal achalasia.
  POEM includes different steps:
  1. Lifting of the esophageal mucosa, with the injection of saline solution, and mucosal incision on the esophageal body (approximately 12 or 7 cm above the esophagogastric junction, for about 1-2cm)
  2. Advance of the endoscope into the submucosa, repeated submucosal injection and dissection of a submucosal tunnel into the distal esophagus up to 3 cm into the gastric wall.
  3. Myotomy of the distal esophagus, cardia and gastric wall, starting 3 cm below the mucosal incision
  4. After the completion of myotomy, and check for mucosal integrity, the mucosal incision is closed using endoscopic clips

SUMMARY:
Per-Oral Endoscopic Myotomy (POEM) is increasingly used for the treatment of achalasia. In published series, a 12cm-POEM is usually performed. Surgical myotomy is typically shorter (8cm). The clinical efficacy of both procedure is comparable.

This study intends to investigate if clinical outcomes of POEM depends on the length of esophageal myotomy, in patients with classic-type achalasia (type I and type II according to Chicago Classification)

DETAILED DESCRIPTION:
Peroral Endoscopic Myotomy myotomy (POEM) has been recently introduced for treatment of achalasia, based on technical developments from NOTES (natural orifice translumenal surgery). The technique includes the incision of the mucosa in the esophageal body, the submucosal dissection of the distal esophagus and the creation of a submucosal tunnel in the distal esophagus and proximal gastric body, and the esophageal myotomy. The procedure is performed transorally, using a flexible endoscope.

In published series, a 12cm-POEM is usually performed. Surgical myotomy is typically shorter, being protracted for about 8cm. The clinical efficacy of POEM and surgical myotomy is more likely to be similar according to the most recent published series.

In this randomized controlled trial (non-inferiority trial) we evaluate the outcomes of POEM according to the length of the esophageal myotomy.

Patients with type I and II achalasia will be randomly assigned to one of the two groups, long--myotomy (LM) and short--myotomy (SM).

Patients in the LM-group will receive a 12cm-long POEM (including 3cm on the stomach); in the SM-group patients will undergo a POEM extended for 7 cm (including 3cm on the stomach).

During follow-up, High Resolution Manometry (HRM), Esophageal pH-monitoring study and Esophagogastroduodenoscopy (EGD) will be regularly performed and symptoms assessed with the use of the Eckardt score (ECKs).

The main hypothesis is that the results of a SM are not inferior to the results of a LM. Calculated sample size is 200 patients

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of achalasia (type I and II)
2. Age > 18
3. Signed informed consent
4. Patient accepts to undergo scheduled follow-up after POEM
5. Eckardt score > 3
6. ASA I-II-III

Exclusion Criteria:

1. Prior surgical treatment of achalasia (previous endoscopic balloon dilation or botox injection ARE NOT exclusion criteria)
2. Pregnancy or nursing
3. Current alcohol or drug addiction.
4. Mentally retarded or emotionally unstable, or exhibits psychological characteristics which, in the opinion of the investigator make the subject a poor candidate for this study.
5. Severe congenital or acquired coagulopathy or INR > 1.6
6. Participating in another ongoing clinical trial in which concomitant diagnosis or therapeutic intervention would adversely affect the integrity of the clinical trial.
7. Hepatic cirrhosis w/ or w/o portal hypertension w/ or w/o esophageal varices
8. Eosinophilic esophagitis or Barrett Esophagus
9. Esophageal Strictures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-06-06 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of a Short-POEM compared to a Long-POEM | 2 years
  Treatment success, defined as an Eckard score ≤ 3.
  The Eckardt score is a clinical score for evaluating the severity of achalasia-related symptoms. Eckardt score varies between 0 and 12.
  Questions are asked about the frequency of dysphagia, regurgitation and retrosternal pressure sensation. Depending on whether any of these symptom occurrs, never, occasionally, daily or with each meal, a symptom score between 0 and 3 is applied. In addition a symptom score of 0-3 is assigned to the degree of weight loss (0 - No weight loss; 1 - weight loss < 5Kg, 2 - weight loss between 5 and 10Kg, 3- weight loss > 10Kg).
  Each symptom score (dysphagia, regurgitation, retrosternal pressure, and wieight loss) is summed to the other. Thus, a completely asymptomatic patient has a score of 0 and the most severely affected patient had a maximum score of 12.

SECONDARY OUTCOMES:
Basal Lower Esophageal Sphincter (LES) pressure | Before POEM, 6 months and 2 years after the procedure
  Basal LES pressure on esophageal manometry after Short-POEM compared to Long-POEM
4-second Integrated Relaxation Pressure (4sIRP) | Before POEM, 6 months and 2 years after the procedure
  4sIRP on esophageal manometry after Short-POEM compared to Long-POEM
Side effects and complications | Baseline to 2 years
  Incidence of side effect and complications after Short-POEM compared to Long-POEM
Gastro-Esophageal Reflux (GER) symptom assessment | baseline, 6 months and 2 years after POEM
  GerdQ questionnaire will be used to evaluate and compare Gastoesophageal reflux symptoms in the two groups.
  GerdQ is a 6-item, validated, easy to use questionnaire. The GerdQ questionnaire asks patients to score the number of days with symptoms and use of over-the-counter (OTC) medications during the previous 7 days. It uses a four graded Likert scale (0-3) to score the frequency of four positive predictors of GERD (heartburn, regurgitation, sleep disturbance due to reflux symptoms or use of over-the-counter (OTC) medications for reflux symptoms) and a reversed Likert scale (3-0) for two negative predictors of GERD (epigastric pain and nausea) giving a total GerdQ score range of 0-18. The sleep disturbance and use of OTC medication are also used for assessment of the impact of GERD, giving a separate 'impact score' ranging from 0 to 6
Esophageal pH-monitoring study | 6 months after POEM
  patients will undergo esophageal pH-monitoring study during the follow-up. DeMeester score will be used for the diagnosis of GERD.
  DeMeester score is a composite score based on 6 parameters (scored in comparison to mean values in normal subjects for each category below):
  Supine reflux, Upright reflux, Total reflux, Number of episodes, Number of episodes longer than 5 min, Longest episode. A score of >14.72 shows significant reflux.
  Prevalence of GERD will be compared in the two study groups
Operating time | During the endoscopic procedure
  The duration of the endoscopic procedures for each patients will be calculated, in minutes, since the mucosal incision until the endoscopic closure of the mucosal entry with the last endoscopic clip.
  The average duration of the procedure in the Short-POEM group will be compared wth the dureation of the procedures in the Long-POEM-groups
Quality of life | baseline, 6 months and 2 years
  Improvement of quality of life after Short-POEM compared to Long-POEM, assessed by using the SF-36 questionnaires' scores
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Familiari P, Borrelli de Andreis F, Landi R, Mangiola F, Boskoski I, Tringali A, Perri V, Costamagna G. Long versus short peroral endoscopic myotomy for the treatment of achalasia: results of a non-inferiority randomised controlled trial. Gut. 2023 Aug;72(8):1442-1450. doi: 10.1136/gutjnl-2021-325579. Epub 2023 Apr 18. PMID 37072180